CLINICAL TRIAL: NCT07366593
Title: Relationship Between Immune Profile and Respiratory Parameters in Down Syndrome Children With Acute Pneumonia: Pre-Intervention Analysis
Brief Title: Immune Profile and Respiratory Parameters in Down Syndrome Children With Acute Pneumonia: Pre-Intervention Analysis
Status: Recruiting | Type: Observational
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Abdelkhalek, assistance professor, Badr University
Other Study IDs: Down Syndrome Children
Record Dates: First submitted 2026-01-13; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome
Keywords: Down Syndrome, pneumonia, immune, oxygen saturation
MeSH Terms: conditions — Down Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pearson or Spearman correlations were used to assess relationships between immune and respiratory variables, and with age — Baseline serum IgG, IgA, IgM (nephelometry), total WBC count (automated analyzer), RR (manual count), and SaO2 (pulse oximetry) were measured. Pearson or Spearman correlations were used to assess relationships between immune and respiratory variables, and with age.

SUMMARY:
Baseline serum IgG, IgA, IgM (nephelometry), total WBC count (automated analyzer), RR (manual count), and SaO2 (pulse oximetry) were measured. Pearson or Spearman correlations were used to assess relationships between immune and respiratory variables, and with age

DETAILED DESCRIPTION:
descriptive, cross-sectional study analyzed baseline data from 40 children with DS and acute pneumonia enrolled prior to intervention in a larger trial. Baseline serum IgG, IgA, IgM (nephelometry), total WBC count (automated analyzer), RR (manual count), and SaO2 (pulse oximetry) were measured. Pearson or Spearman correlations were used to assess relationships between immune and respiratory variables, and with age.

ELIGIBILITY:
Inclusion Criteria:

* Down Syndrome with acute bronchopneumonia
* sufficient cognitive ability

Exclusion Criteria:

* severe congenital heart defects
* primary immunodeficiencies

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Data collection occurred at the inpatient pediatric ward of King Abdulaziz University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
serum IgG, IgA, IgM | Upon enrollment and prior to any intervention baseline data were collected
  Immunoglobulins: Concentrations of IgG(mg/dl) IgA,(mg/dl) and IgM (mg/dl) were determined from serum using an automated nephelometer
Respiratory Rate | Upon enrollment and prior to any intervention baseline data were collected
  Respiratory rate (breaths/minute) was determined by direct observation and counting of chest wall movements over one full minute
Arterial Oxygen Saturation (SaO2) | Upon enrollment and prior to any intervention baseline data were collected
  Peripheral oxygen saturation (%) was measured non-invasively via pulse oximetry
White Blood Cell count | Upon enrollment and prior to any intervention baseline data were collected
  Total WBC count (thousands/mm³) was measured from a whole blood sample using an ADVIA 120 automated hematology analyzer

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Badr university, Cairo
  - Mona Mohamed Abdelkhalek, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet determined whether individual participant data will be shared. Any future decision will depend on institutional policies, ethical considerations, and applicable data protection regulations."